CLINICAL TRIAL: NCT06646549
Title: The Association of Insomnia With Fatigue and Mood in Postmenopausal Osteoporosis
Brief Title: Insomnia in Postmenopausal Osteoporosis
Status: Completed | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: Beylikdüzüstateh4
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Aim of the study was to determine the presence of sleep problems in postmenopausal osteoporosis patients and to examine the relationship between the severity of insomnia and mood and fatigue. Pain, sleep problems, depression, anxiety, and fatigue were assessed using appropriate scales

DETAILED DESCRIPTION:
The research was planned as a clinical cross-sectional study. Two hundred women, aged between 50-75 years, who were diagnosed with postmenopausal osteoporosis and followed up in the outpatient clinics of Beylikdüzü State Hospital and Istanbul Physical Medicine and Rehabilitation Training and Research Hospital between May 19, 2024, and June 19, 2024, were included. Sociodemographic data such as gender, height, weight, body mass index, educational status, and occupation were recorded. The date of osteoporosis diagnosis, history of falls within the last 6 months, presence of fractures due to low-energy trauma, osteoporosis treatment, medications used, and comorbidities were questioned. The presence and location of pain were asked, and if pain was present, its intensity was determined using the Visual Analog Scale. Calcium and vitamin D levels from the last 3 months were recorded. The patient's sleep problems were assessed using the Insomnia Severity Index. Subsequently, the patient's current depression and anxiety-related symptoms were measured using the Hospital Anxiety and Depression Scale (HADS), and the fatigue level was assessed with the Fatigue Severity Scale (FSS).

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with postmenopausal osteoporosis.
* Patients who agreed to participate in the study.
* Age range between 50-75 years.

Exclusion Criteria:

* Presence of fibromyalgia.
* Chronic fatigue syndrome.
* Chronic decompensated cardiac, renal, or hepatic failure.
* Known psychiatric disorders.
* Rheumatological diseases.
* Presence of other known neurological diseases.
* Use of medications that enhance physical performance or alleviate fatigue.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with postmenopausal osteoporosis were included in the study.
Study Population: Women diagnosed with postmenopausal osteoporosis.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-05-19 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | 0 day
  The Insomnia Severity Index (ISI) is a widely used, validated tool designed to assess the nature, severity, and impact of insomnia. It is a brief, self-report questionnaire consisting of seven items that evaluate various aspects of insomnia, including difficulties falling asleep, staying asleep, waking up too early, satisfaction with sleep, interference with daily functioning, noticeable impairments, and distress caused by sleep problems.The score ranges from 0 to 28. As the score increases, the severity of insomnia worsens.

SECONDARY OUTCOMES:
Fatigue Severity Scale | 0 day
  The Fatigue Severity Scale (FSS) is a commonly used self-report tool designed to assess the impact and severity of fatigue on an individual's daily life. It consists of nine statements related to fatigue and its influence on physical and mental activities, motivation, and social functioning. Each statement is rated on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree), with higher scores indicating greater fatigue severity.The score ranges from 9 to 63. A higher score indicates more severe fatigue, meaning the condition worsens with increasing scores.
Hospital Anxiety and Depression Scale | 0 day
  The Hospital Anxiety and Depression Scale (HADS) is a widely used screening tool designed to identify symptoms of anxiety and depression in individuals, particularly in non-psychiatric hospital settings. It was developed to avoid reliance on physical symptoms, which may be more related to a person's medical condition rather than to anxiety or depression.Each subscale (anxiety and depression) ranges from 0 to 21. As the score increases, the severity of anxiety or depression worsens.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Şirin Ahısha, MD, Principal Investigator — Beylikdüzü State Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Beylikdüzü State Hospital, Istanbul, Beylikdüzü
  - Beylikdüzü State Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No